CLINICAL TRIAL: NCT06655272
Title: OM 85 to Prevent Respiratory Infections in Older At Risk Patients
Acronym: OM85OLDER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Collaborators: OM Pharma SA (Industry)
Responsible Party: Principal Investigator, Raffaele Antonelli Incalzi, Professor, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 23892; 2024-513592-41-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Tract Infections (RTI)
Keywords: Older people; Nursing home; Bacterial lysate
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Broncho-Vaxom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Bacterial lysate p.o. administered for two three-months cycles.
  Interventions: Drug: Bacterial Lysate
- Control (Placebo Comparator): Matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bacterial Lysate — Administration p.o. for 10 days per month for 3 months, two consecutive cycles.
  Arms: Intervention
Drug: Placebo — Matching placebo.
  Arms: Control

SUMMARY:
People living in NH are at higher risk of respiratory infections compared to their counterpart living in the community. Products obtained from dead bacteria ("bacterial lysate") can be used to boost immune system and may reduce the risk of respiratory infections. Very little information is available on the effect of these substances in older people. This study will evaluate the efficacy of a bacterial lysate in reducing the incidence of lower respiratory tract infections in older people living in nursing homes. The study will include a treatment arm, in which participants will received the lysate, and a control arm in which participants will received a matching placebo (i.e., a pill that has the same appearance of the lysate but does not contain the lysate itself).

DETAILED DESCRIPTION:
OM 85 (lyophilized bacterial lysate) proved effective in increasing the immune response against bacteria in animal models. Furthermore, its use was shown to be associated with lower incidence of RTIs in children and at risk adults. However, there is a paucity of information about OM 85 efficacy in the elderly, i.e., in a population which, due to immunosenescence and multimorbidity, might have a distinctive response to this immunostimulating strategy. Indeed, the only study properly designed for a geriatric population is a randomized controlled trial on 290 people over-65 with chronic bronchitis and frequent exacerbations; here, a significant decrease in the incidence of acute bronchitis was observed in the OM 85 group over 6 months (Orcel B et al. Eur Respir J, 1994, 7, 446-452). However, this population seems poorly representative of the average older population at risk of RTI. Indeed, chronic diseases like congestive heart failure and chronic renal failure qualified as exclusion criteria. Furthermore, a history of at least 4 episodes of acute bronchitis treated with antibiotics in the 6-month reference period of the previous year were requested for the enrollment. Thus, the study population is unlikely to reflect the profile of risk of the elderly and frail population, which is characterized by a high prevalence of chronic diseases, but not by such a high incidence of respiratory infections. Indeed, even in severe COPD the frequency of exacerbations rarely exceeds 2 yearly and is rapidly declining (Andreas et al. Respiratory Research (2019) 20:186). Geriatric patients are variably represented in other studies which proved the efficacy of OM 85 in adult populations with COPD or chronic bronchitis. Twelve studies met the quality criteria to be eligible for a recently published meta-analysis (Huang Y, Pei Y, Qian Y, Yao Z, Chen C, Du J, Shi M, and Zhou T, 2022. A meta-analysis on the efficacy and safety of bacterial lysates in chronic obstructive pulmonary disease. Front. Med. 9:877124. doi: 10.3389/fmed.2022.877124). However, elderly patients and especially those over 75, the most vulnerable to respiratory infections, were a minority of probands. Furthermore, the selection criteria pointed at COPD as the main disease in the vast majority of the studies. IMP has never been tested in an older population with a heavy burden of multimorbility and frailty and a high risk of RTI, I e in the population most likely to benefit from it. Accordingly, this trial is expected to clarify what previous studies could not because they were not designed to study this kind of population, and only sparse and partial information could be derived by picking selected patients from the study populations. Furthermore, all our patients will receive the recommended vaccines, and this will allow test IMP in a framework free from confounding by heterogeneity in vaccine policy.

Primary objective:

To evaluate whether and to which extent OM85 compared with placebo is able to reduce respiratory tract infections (RTIs) over a 12-month period in a population of subjects aged 75 years and older, residing in nursing homes, and with a history of at least two RTIs in the 12 months prior to enrollment.

Secondary objectives:

To verify whether the rate of hospital admissions and emergency department visits due to RTI decreases from the previous year differently in the OM 85 group compared with placebo.

Evaluate the number of antibiotic prescriptions between the two groups (OM 85 and placebo) during the 12-month study period.

Describe the demographic, clinical and functional characteristics of patients with higher RTI numbers.

Evaluate the incidence of treatment-emergent adverse events (TEAEs).

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years or older
* At least 2 RTIs in the year prior to enrollment
* Patients must have been residing in nursing homes for at least 6 months and have an estimated length of stay in nursing homes of at least 6 months by their treating physician.
* Signed informed consent. If participants are unable to provide informed consent due to cognitive impairment, consent will be provided by a legally recognized representative or trustee of the patient (pursuant to Article 4 of Law No. 219 of December 22, 2017).
* Have a life expectancy of at least one year in the judgment of their treating physician.

Exclusion Criteria:

* Patients with known allergy or previous intolerance to any component (including the excipient) of the study drug
* Patients with active neoplasia and prognosis of less than one year
* Patients with previous organ transplantation
* Patients treated with prohibited drugs (see Table 1) in the 3 months prior to the start of the study
* Patients who have taken bacterial lysates in the 6 months prior to enrollment or are currently using them
* Patients regularly treated with oral corticosteroids
* Patients unable to follow instructions and unreliable patients (including patients with alcoholism or patients unwilling to give informed consent or comply with protocol requirements)
* Patients with any other clinical condition that, in the opinion of the investigator, would not allow completion of the protocol and safe administration of the study drugs

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of lower respiratory tract infections. | 12 months
  New cases of clinically-diagnosed lower respiratory tract infections

SECONDARY OUTCOMES:
Rate of hospitalizations and emergency room admissions | 12 months
  Rate of hospitalizations and emergency room admissions due to respiratory tract infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Campus Bio-Medico, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No